CLINICAL TRIAL: NCT05697406
Title: Hyperpolarized 13-C Pyruvate MRI Surveillance of Multiple Cancers
Brief Title: HP Pyruvate MRI in Cancers
Acronym: HC-MRI
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Vikas Kundra, Chief of Oncologic Imaging, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HP-00101177
Record Dates: First submitted 2023-01-06; First posted 2023-01-25 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Image; Warburg Effect; Tumors
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants will be evaluated pre and post hyperpolarized 13-C pyruvate injection for change in pyruvate signal compared to background.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental (Experimental): Participants will receive an injection of 250 mM of hyperpolarized 13-C pyruvate intravenously after standard of care imaging sequences are performed. Then participants will undergo HP-MR imaging.
  Interventions: Drug: Hyperpolarized 13C-Pyruvate

INTERVENTIONS:
Drug: Hyperpolarized 13C-Pyruvate — Imaging tumors pre and post administration of hyperpolarized 13-C pyruvate injection.

SUMMARY:
Many human diseases are characterized by their ability to alter existing metabolic pathways and interrupt cellular processes. Cancer exploits the Warburg effect and utilizes greater glucose than normal cells and within this process uses anaerobic respiration, leading to increased conversion of pyruvate to lactate. This can be exploited by hyperpolarized imaging. Hyperpolarized 13C MRI imaging is an approach that utilizes a stable isotope of Carbon (13C) linked to pyruvate. MRI spectroscopy is used in conjunction with hyperpolarized 13C pyruvate in order to temporally detect pyruvate and its conversion to lactate in-vivo, in order to visualize downstream metabolic (glycolytic) activity secondary to the Warburg effect, which should be useful in detecting and characterizing tumors of various types. Hyperpolarized 13C pyruvate MR imaging has not been tested in most cancers. In this preliminary survey, we will test the hypothesis that hyperpolarized 13C pyruvate MR imaging can be used to image various cancers.

DETAILED DESCRIPTION:
Most cancers exhibit the Warburg effect, which involves synthesis of lactate via glycolytic pathways. The present method of using 18F-FDG to image metabolic events only evaluates early glycolysis and does not investigate late glycolytic effects which can be examined by 13C pyruvate. The ability to detect cancer using 13C pyruvate has been shown using ovarian cancer models and in the prostate in humans, however its utility in other tumors needs clarification. Because cancers of various types affect metabolic pathways, it is necessary to improve imaging techniques to better investigate downstream metabolism. Many studies have shown that there are higher lactate levels in cancer tissue and higher levels of glycolysis. 13C pyruvate imaging takes advantage of these pathways by imaging the tumors while undergoing pyruvate to lactate conversion . From this modality, a three dimensional visualization of the tumor and metabolic products created by the pyruvate can be investigated.

ELIGIBILITY:
Inclusion Criteria:

Clinical tumor diagnosis

Patients with pre-existing MR imaging appointments

Must be able to undergo MR

Exclusion Criteria:

No tumor diagnosis

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Pyruvate to Lactate Conversion | 18-36 months
  Imaging Quality, KpL

SECONDARY OUTCOMES:
SNR | 12-42 months
  Signal to Noise Ratio, dB
CNR | 12-42 months
  Contrast to Noise

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Di Lorenzo R, Bernardi M, Genedani S, Zirilli E, Grossi G, Guaraldi GP, Bertolini A. Acute alkalosis, but not acute hypocalcemia, increases panic behavior in an animal model. Physiol Behav. 1987;41(4):357-60. doi: 10.1016/0031-9384(87)90401-x. PMID 2829248
- [Background] Roberts GE, Heeley AF. Tryptophan metabolism in psychotic children. Dev Med Child Neurol. 1968 Oct;10(5):681. No abstract available. PMID 5708291
- [Background] Wang ZJ, Ohliger MA, Larson PEZ, Gordon JW, Bok RA, Slater J, Villanueva-Meyer JE, Hess CP, Kurhanewicz J, Vigneron DB. Hyperpolarized 13C MRI: State of the Art and Future Directions. Radiology. 2019 May;291(2):273-284. doi: 10.1148/radiol.2019182391. Epub 2019 Mar 5. PMID 30835184